CLINICAL TRIAL: NCT03314454
Title: Alcohol Use and Mental Health - Pilot Test of Video-assisted Drinking Topography
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This was an internally-funded pilot and priority had to be given to grant-funded projects.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB201700455
Record Dates: First submitted 2017-10-04; First posted 2017-10-19 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Beer

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are aware of the interventions, but are not aware of the assigned arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Elevated Mental Status (Active Comparator): Elevated score on Patient Health Questionnaire
  Interventions: Drug: Beer; Device: Videotaped drinking session
- Non-elevated depressed mood (Active Comparator): Lower score on Patient Health Questionnaire
  Interventions: Drug: Beer; Device: Videotaped drinking session
- Social Drinking status (Active Comparator): The social drinker group will be those who consume alcohol regularly but with infrequent heavy drinking days.
  Interventions: Drug: Beer; Device: Videotaped drinking session
- Heavy drinker status (Active Comparator): The heavy drinker group will be those who consume alcohol regularly with frequent heavy drinking days.
  Interventions: Drug: Beer; Device: Videotaped drinking session

INTERVENTIONS:
Drug: Beer — Common brands beer with similar calorie (125-150) and alcohol level (approximately 4.5% ABV)
Device: Videotaped drinking session — Video-assisted alcohol topography to explore its utility as an indicator of alcohol use disorder
  Other Names: video-assisted topography

SUMMARY:
The overall goal is to pilot test and establish a procedure for video-assisted alcohol topography and explore its utility as an indicator of alcohol use disorder. There are 4 phases to this study: 1) pre-screening by phone; 2) in-person screening appointment; 3) the first alcohol drinking session with videotaping; and 4) follow-up appointment for retest.

DETAILED DESCRIPTION:
Alcohol use especially high-risk drinking remains a serious public health concern. Recent calls for "precision intervention" require more in-depth understanding of drinking behavioral patterns for more individualized treatment. Currently, alcohol research has relied on self-reported questionnaire or biomarkers to measure alcohol use. However, self-reports are often subjected to social desirability bias or recall errors; whereas biomarkers are prone to measurement errors, confounders for false positives, and individual variations in alcohol metabolism. There is need for an objective, reliable, and nonintrusive way to measure alcohol use with high ecological validity.

Topography can provide objective measures of consumption behavior patterns in fine grained detail. While it has been widely used in tobacco research, alcohol topography has not been well-studied. Smoking topography has been shown to provide indicative information for nicotine dependence. The investigators hypothesize that alcohol topography can also be used as an objective measure indicative of alcohol use disorder. In this project, the investigators propose to conduct a video-assisted drinking topographical study. The main objectives of this study include: (1) characterize drinking behavioral patterns by converting videotaped drinking episodes into various drinking related parameters (e.g., sipping frequency, sipping interval, sipping duration, rest duration, sipping amount, and etc.); (2) compare drinking behavioral patterns across groups defined by drinking status (social vs. heavy drinkers) and mental health status (depressed vs. non-depressed); and (3) use advanced nonlinear modeling to quantify the behavioral pattern and to derive potential indicators for alcohol use disorder.

This will be the first study to ever use videotaped topography to analyze alcohol drinking behavioral pattern using a quantum model and link it to alcohol use disorder. The study will be conducted in the simulated bar laboratory located in Yon Hall at the University of Florida (UF). Conducting alcohol topography in such a setting greatly enhances ecological validity, further increasing the capacity of this method to capture real life drinking patterns and to potentially detect alcohol use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Be able to read/write English and complete study assessments
* Drink alcohol
* Healthy adults reporting alcohol consumption in the past 30 days
* Not currently seeking treatment for substance use
* Willingness to provide urine drug screening

Exclusion Criteria:

* Test positive on a urine test for use of certain illegal drugs
* Undergraduate student enrolled at the University of Florida
* Graduate students from the College of Health and Human Performance at the University of Florida
* Pregnant, or currently breast feeding

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Leeman, PhD, Principal Investigator — University of Florida
Locations (1):
- EDGE Laboratory, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We did not get far enough along with recruitment for this pilot study to recruit social drinkers, nor individuals with elevated mental status thus all participants recruited were considered to have heavy drinker status with non-elevated depressed mood, thus precluding comparisons between these groups.
Pre-assignment Details: As explained in recruitment details, enrollment for this pilot study ended early before social drinkers or participants with elevated mental status could be recruited, thus precluding group comparisons.
Groups:
- Single Arm: Heavy Drinking Only With Elevated and Non-elevated Depressed Mood: We terminated this study early with only 10 of the projected 40 participants completing an alcohol administration laboratory session. We terminated the study before we could recruit social drinkers or participants with elevated mental status. For other classifications, subgroup sizes are too small for these results to have any meaning, thus we opted to present these results descriptively as a single group including only those with heavy drinking and both elevated and non-elevated depressed mood.
Period: Overall Study
Arm/Group | Single Arm: Heavy Drinking Only With Elevated and Non-elevated Depressed Mood
Started | 11
Completed | 10
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: We ended this study early, with only 10 of the projected 40 participants completing an alcohol administration laboratory session, before we could recruit social drinkers or participants with elevated mental status. For other classifications, subgroup sizes are too small for these results to have any meaning, thus we opted to present these results descriptively as a single group.
Groups:
- Study Sample: We ended this study early, with only 10 of the projected 40 participants completing an alcohol administration laboratory session, before we could recruit social drinkers or participants with elevated mental status. For other classifications, subgroup sizes are too small for these results to have any meaning, thus we opted to present these results descriptively as a single group.
Arm/Group | Study Sample
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants] — Age range recruited for study
  Participants
    <=18 years | 0
    Between 18 and 65 years | 10
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Self-reported sex at birth
  Participants
    Female | 4
    Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: White, non-Hispanic | 7
  Race/ethnicity: Black, non-Hispanic | 2
  Race/ethnicity: Asian, non-Hispanic | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Topography: Sip Frequency
Description: To explore the potential of using alcohol topography as a noninvasive objective measure of alcohol drinking behavior and the possibility of using the identified behavioral pattern as an indicator for alcohol use disorder. We operationalized alcohol topography in several ways including the present measure: mean number of sips per alcoholic drink
Time Frame: 60 days (from phone screening to follow-up retest)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: sips per drink
Arm/Group | Study Sample
Number analyzed (Participants) | 10
sips per drink | 14.67 (7.57)

2. Primary Outcome: Alcohol Topography: Sip Interval
Description: To explore the potential of using alcohol topography as a noninvasive objective measure of alcohol drinking behavior and the possibility of using the identified behavioral pattern as an indicator for alcohol use disorder. We operationalized alcohol topography in several ways including the present measure: mean interval between sips
Time Frame: 60 days (from phone screening to follow-up retest)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Study Sample
Number analyzed (Participants) | 10
minutes | 1.46 (1.03)

3. Primary Outcome: Alcohol Topography: Sip Duration
Description: To explore the potential of using alcohol topography as a noninvasive objective measure of alcohol drinking behavior and the possibility of using the identified behavioral pattern as an indicator for alcohol use disorder. We operationalized alcohol topography in several ways including the present measure: mean sip duration
Time Frame: 60 days (from phone screening to follow-up retest)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Study Sample
Number analyzed (Participants) | 10
seconds | 2.01 (0.43)

4. Primary Outcome: Alcohol Topography: Sip Amount.
Description: To explore the potential of using alcohol topography as a noninvasive objective measure of alcohol drinking behavior and the possibility of using the identified behavioral pattern as an indicator for alcohol use disorder. We operationalized alcohol topography in multiple ways including the current measure: mean amount of beer consumed per sip
Time Frame: 60 days (from phone screening to follow-up retest)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: grams per sip
Arm/Group | Study Sample
Number analyzed (Participants) | 10
grams per sip | 32.35 (19.84)

ADVERSE EVENTS:
Time Frame: 16 months
Description: We ended this study early, with only 10 of the projected 40 participants completing an alcohol administration laboratory session, before we could recruit social drinkers or participants with elevated mental status. For other classifications, subgroup sizes are too small for these results to have any meaning, thus we opted to present adverse events (of which there were none) among the full sample only
Groups:
- Study Sample: We ended this study early, with only 10 of the projected 40 participants completing an alcohol administration laboratory session, before we could recruit social drinkers or participants with elevated mental status. For other classifications, subgroup sizes are too small for these results to have any meaning, thus we opted to present adverse events (of which there were none) among the full sample only
Arm/Group | Study Sample
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT03314454/Prot_SAP_001.pdf